CLINICAL TRIAL: NCT00325182
Title: The Effects of Levetiracetam on Alcohol Dependent Subjects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-23008
Record Dates: First submitted 2006-05-11; First posted 2006-05-12 (Estimated); Last update posted 2017-03-15 (Actual); Status verified 2007-04

CONDITIONS: Alcoholism
Keywords: Alcoholism
MeSH Terms: conditions — Alcoholism | interventions — Levetiracetam

ARMS (2):
- Intervention: Levetiracetam (Experimental): Levetiracetam dose schedule Days 1-4 250 mg bid Days 5- 19 500 mg bid Days 20 -70 1000 mg bid Days 71-78 500 mg bid Days 79-85 250 mg bid Days 86-91
  Interventions: Drug: Levetiracetam
- Historical controls (Placebo Comparator): Historical controls from COMBINE study who receive a placebo
  Interventions: Other: Historical controls

INTERVENTIONS:
Drug: Levetiracetam
  Other Names: Keppra
  Arms: Intervention: Levetiracetam
Other: Historical controls
  Arms: Historical controls

SUMMARY:
This study will attempt to examine whether Levetiracetam (Keppra (TM)) can help people with alcohol dependence cut down on their alcohol consumption. In addition, the investigation will assess the effectiveness of Keppra on reducing withdrawal symptoms post alcohol cessation. Matched group of historical controls of alcohol dependent patients receiving placebo will be used for comparison.Based on the mechanism of action of Keppra we hypothesize that it may be effective in promoting abstinence and reducing drinking behavior in alcohol dependent patients.

DETAILED DESCRIPTION:
Alcoholism is a chronic disease with numerous psychological, social and medical consequences. Alcohol use disorders are one of the most prevalent psychiatric disorders in general population in the US. Alcoholism not only disrupts an individual's life, health and ability to function in the society, has tremendous impact on families and communities, but also is associated with enormous economic cost for society. The medical and social impact of alcoholism can be reduced via effective treatments. Although medical, psychological and social approaches have demonstrated some efficacy, no specific method has consistently shown superiority. Similarly, currently available pharmacological treatments for alcohol use disorders are associated with moderate efficacy, indicating that further efforts are required to develop novel interventions.

The rewarding effects of alcohol are at least partially mediated via dopamine pathways that originate in the ventral tegmental area and project to the nucleus accumbens. Alcohol through its effects on GABA receptor activity decreases the inhibitory effect of GABA on the dopaminergic neurons in ventral tegmental area and therefore facilitates dopamine neurotransmission. Medications that modulate excitatory neurotransmission in the brain (glutamate) and facilitate inhibitory effects of GABA have been shown to be clinically effective in treatment of alcoholism.

Keppra is a novel antiepileptic medication currently approved for treatment of partial onset seizures as an adjunctive agent. It has a unique mechanism of action in that it reduces negative allosteric effects of Zn++ and Beta- carboline in two main inhibitory receptors in the CNS- the GABA A and glycine receptors. These modulators inhibit the influx of chloride though both of these receptor complexes and are therefore considered excitatory mediators. Keppra prevents the negative modulation and promotes chloride flux, thereby, inhibiting neurotransmission.

Limited laboratory work with levetiracetam (Keppra) has shown that the medication can reverse the anxiogenic effect of benzodiazepine withdrawal in mice (Y. Lamberty et al., 2002). Furthermore, Keppra was investigated for its potential to prevent alcohol withdrawal symptoms in mice. In this study levetiracetam dose-dependently prevented spontaneous tremors and handling induced convulsions in alcohol dependent mice. (Y. Lamberty et al., 2002). Based on the mechanism of action of Keppra we hypothesize that it may be effective in promoting abstinence and reducing drinking behavior in alcohol dependent patients.

ELIGIBILITY:
Inclusion Criteria:

* DSM IV TR Diagnosis of Alcohol Dependence
* Male or female age 21-60 years old
* Able to provide informed consent and comprehend study procedures
* Negative urine toxicological screen for narcotics, amphetamines, sedative hypnotics and cannabinoids. The test may be repeated within a week.
* Score of > 8 on Alcohol Use Disorder Identification Test during screening
* Must be suitable for outpatient management
* Express desire to stop drinking or reduce alcohol consumption with possible long-term goal of abstinence.
* Provide contact information for themselves or an alternate contact that the study staff will contact in case of missed appointment.
* Female subjects must be postmenopausal for at least one year, or practicing an effective method of birth control before entry and throughout the study
* Must be able to take oral medications, adhere to regimen and be willing to return for follow up visits
* Must have breath alcohol concentration of no more than 0.025% when signing the informed consent

Exclusion criteria:

* Dependent on or extensive abuse of drugs or substances other than ethanol, nicotine or caffeine
* DSM IV- TR diagnosis of any current Axis I diagnosis other than alcohol, nicotine or caffeine dependence that in the investigator's judgment might require intervention with either pharmacological or non-pharmacological therapy that might interfere with the course of the study
* Receiving inpatient or outpatient treatment for alcohol dependence (with the exception of AA or other self-help groups) within the 4 weeks prior to enrollment
* Subjects with a score of 10 or greater on the CIWA-Ar at visits one and two
* Currently being treated with disulfiram or naltrexone
* Currently being treated with any the following medications: a) Antipsychotic agent [b) Lithium Carbonate c) Anticonvulsant agent d) Hypnotics e) Antianxiety Agents f) Chronic opiate treatment with methadone, laam, buprenorphine; oxycodone, morphine, etc g) Stimulant treatment
* Subjects who are legally mandated to participate in alcohol treatment program
* Subjects who have had a suicide attempt or suicidal ideation within 30 days of the first visit
* Subjects with renal disease
* Subjects with AST and ALT >3 times the upper limit of the normal range during screening. Test may be repeated prior to enrollment. If repeat lab values are all within acceptable ranges subject may continue study participation.
* Major neurological disorder including seizures
* Subjects who are pregnant or lactating
* Subjects known to have clinically significant medical conditions, including, but not limited to: symptomatic CAD or PVD, malignancy or history of malignancy in the last 5 years, pulmonary disorders, endocrinological disorders
* Subjects with prior hypersensitivity to Keppra
* Subjects with history of medically complicated withdrawal from alcohol.
* Subjects who in the opinion of the investigator should not be enrolled in the study because of the precautions, warnings and contraindications outlined in the Keppra package insert
* Subjects with cardiac pacemaker or metal surgical implant

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2006-01 (Actual); Primary Completion 2007-01 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Change in mean number of drinks | Baseline and at 11 weeks
  The primary outcome of this study will be determined by comparing the mean drinks consumed per day at baseline (the month prior to the screening session) compared with the mean drinks per day consumed during week 11 of the treatment period.

SECONDARY OUTCOMES:
Heavy drinks per drinking day | At 13 weeks and last value carries forward approaches
  Mean heavy drinks per drinking day, OCDS scores, MOS-Sleep Scores, and POMS scores.
OCDS scores, MOS-Sleep Scores, and POMS scores. | At 13 weeks and last value carries forward approaches
  Mean OCDS scores, MOS-Sleep Scores, and POMS scores.

CONTACTS AND LOCATIONS:
Overall Officials: Ofra Sarid-Segal, MD, Principal Investigator — Boston University
Locations (1):
- Boston University Dept of Psychiatry Clinical Studies Unit, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No